CLINICAL TRIAL: NCT00312416
Title: Effects of Topical Clonidine vs. Brimonidine on Choroidal Blood Flow and Intraocular Pressure During Isometric Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-121203B
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Ocular Physiology; Regional Blood Flow
Keywords: Choroidal blood flow; Clonidin; Brimonidin
MeSH Terms: interventions — Clonidine; Brimonidine Tartrate

INTERVENTIONS:
Drug: Clonidin
Drug: Brimonidine

SUMMARY:
Brimonidine tartrate is an alpha-2 agonist ocular hypotensive drug that exerts its effect by causing both a decrease in aqueous production and an increase in uveoscleral outflow. It has been proven to reduce increased intraocular pressure in glaucoma and ocular hypertension. As an alpha 2 agonist Brimonidine belongs to the same class of drugs as Clonidine; however, its molecular structure is sufficiently different to make it more selective for the alpha 2 receptor than Clonidine. Unlike Clonidine, Brimonidine does not appear to have an effect on the central nervous system and therefore does not cause sedation or systemic hypotension.

In addition to their known effect of lowering intraocular pressure, alpha 2 adrenoceptor agonists are neuroprotective. It has, however, been shown that Brimonidine is a very potent vasoconstrictor in the ciliary body thus reducing aqueous humor production. Little is, however, known about potential vasoconstrictor effects of Brimonidine in the posterior pole of the eye. This is of clinical importance, because optic nerve head ischemia appears to contribute to glaucoma pathophysiology.

This study is performed to investigate the effects of topical Clonidine vs. topical Brimonidine on choroidal blood flow and intraocular pressure during isometric exercise.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must A et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 Dpt.
* Intraocular pressure between 10 and 18 mmHg.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* History or family history of epilepsy

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2004-02; Study Completion 2004-12

PRIMARY OUTCOMES:
Choroidal pressure-flow relationship

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjäger-Mayrl, M.D., Principal Investigator — Deapartment of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria